CLINICAL TRIAL: NCT01849692
Title: A Prospective, Two-Staged, Single-Masked Study to Evaluate the Effect of ESBA1008 Applied by Microvolume Injection or Infusion in Subjects With Exudative Age-Related Macular Degeneration
Brief Title: ESBA1008 Microvolume Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-13-001
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-01

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Exudative Age-Related Macular Degeneration; Wet AMD; Choroidal neovascularization (CNV); Vascular endothelial growth factor (VEGF)
MeSH Terms: conditions — Choroidal Neovascularization | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ESBA1008 1.2 mg/10 μL (Experimental): Cohort 1: One intravitreal injection on Day 0, followed by one intravitreal (IVT) injection of ESBA1008 6 mg/50 μL on Day 28
  Interventions: Drug: ESBA1008 solution
- ESBA1008 1 mg/8.3 μL (Experimental): Cohort 2: One intravitreal infusion on Day 0, followed by one intravitreal injection of ESBA1008 6 mg/50 μL on Day 28
  Interventions: Drug: ESBA1008 solution
- ESBA1008 0.6 mg/10 μL (Experimental): Cohort 3: One intravitreal injection on Day 0, followed by one intravitreal injection of ESBA1008 6 mg/50 μL on Day 28
  Interventions: Drug: ESBA1008 solution
- ESBA1008 0.5 mg/8.3 μL (Experimental): Cohort 4: One intravitreal infusion on Day 0, followed by one intravitreal injection of ESBA1008 6 mg/50 μL on Day 28
  Interventions: Drug: ESBA1008 solution
- Ranibizumab 0.5 mg in 50 μL (Active Comparator): Cohorts 1-4: One intravitreal injection on Day 0, followed by another intravitreal injection on Day 28
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: ESBA1008 solution — Intravitreal injection or infusion
  Arms: ESBA1008 0.5 mg/8.3 μL; ESBA1008 0.6 mg/10 μL; ESBA1008 1 mg/8.3 μL; ESBA1008 1.2 mg/10 μL
Drug: Ranibizumab — Intravitreal injection
  Other Names: LUCENTIS®
  Arms: Ranibizumab 0.5 mg in 50 μL

SUMMARY:
The purpose of this study is to demonstrate a treatment effect of ESBA1008 applied as a microvolume injection or infusion on retinal function and morphology in subjects with exudative age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
This 4-cohort study was conducted in 2 stages. Stage 1 consisted out of 2 Cohorts. In each cohort subjects were randomized 10:3 to either receive ESBA1008 (Cohort 1 : 2 injections, Cohort 2 : 1 infusion and 1 injection) or 2 Lucentis injections. Stage 2 was conducted similarly with a different dosing level for ESBA1008 (Cohort 3 and 4). Subjects had follow-up visits at Day 7 and Day 14. All cohorts receiving ESBA1008 on Day 0 also received ESBA1008 6mg/50 μL via injection on Day 28. After the Day 28 visit (all cohorts), subjects returned for follow up visits at Day 42 and Day 56.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent document;
* Able to make the required study visits and follow instructions;
* Age-related macular degeneration in the study eye;
* Visual acuity within protocol-specified range;
* 340 μm minimal central subfield thickness (CSFT; Spectralis Equivalent)
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Both eyes: Any active infection or inflammation;
* Study eye: Any treatment for exudative age-related macular degeneration (AMD) other than vitamin supplements;
* Study eye: Any current or history of macular or retinal disease;
* Study eye: Any concurrent intraocular condition such as cataract or diabetic retinopathy that, in the opinion of the Investigator, could either require medical or surgical intervention during the course of the study to prevent or treat visual loss;
* Study eye: Other ocular conditions or diseases that, in the opinion of the Investigator, could compromise visual acuity;
* Study Eye: Uncontrolled glaucoma;
* History of a medical condition that, in the opinion of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product;
* Women of childbearing potential who are lactating, pregnant, planning to become pregnant, or not using adequate birth control methods for the duration of the study;
* Intraocular surgery within 3 months of baseline;
* Study eye: Any history or current evidence of retinal angiomatous proliferation (RAP) lesions based on clinical exam;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Group Leader, GCRA, Pharma, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 investigational centers located in the US, Australia, and the Dominican Republic.
Pre-assignment Details: Of the 107 enrolled, 55 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized participants (52).
Groups:
- Cohort 1 - ESBA: ESBA1008 solution Day 0 (1.2 mg) and Day 28 (6 mg)
- Cohort 1 - Ranibizumab; Cohort 2 - Ranibizumab; Cohort 3 - Ranibizumab; Cohort 4 - Ranibizumab: Ranibizumab 0.5 mg injection, Day 0 and Day 28
- Cohort 2 - ESBA: ESBA1008 solution Day 0 (1 mg) and Day 28 (6 mg)
- Cohort 3 - ESBA: ESBA1008 solution Day 0 (0.6 mg) and Day 28 (6 mg)
- Cohort 4 - ESBA: ESBA1008 solution Day 0 (0.5 mg) and Day 28 (6 mg)
Period: Overall Study
Arm/Group | Cohort 1 - ESBA | Cohort 1 - Ranibizumab | Cohort 2 - ESBA | Cohort 2 - Ranibizumab | Cohort 3 - ESBA | Cohort 3 - Ranibizumab | Cohort 4 - ESBA | Cohort 4 - Ranibizumab
Started | 10 | 3 | 10 | 3 | 10 | 3 | 10 | 3
Completed | 10 | 3 | 10 | 3 | 10 | 3 | 10 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all subjects who were randomized, received the initial injection or infusion, and had a baseline value and at least 1 postbaseline measurement for the period up to Day 28 for the primary efficacy variables (BCVA and/or CSFT). Here, "n" is the number of subjects in each cohort for each arm group, respectively.
Groups:
- ESBA: All subjects who were treated with ESBA1008.
- LUCENTIS: All subjects who were treated with LUCENTIS.
- Total: Total of all reporting groups
Arm/Group | ESBA | LUCENTIS | Total
Number analyzed (Participants) | 40 | 12 | 52
Age, Continuous [Mean (Standard Deviation); unit: years]
  Cohort 1, n=10, 3 | 77.5 (3.6) | 78.3 (7.2) | 77.7 (4.3)
  Cohort 2, n=10, 3 | 73.6 (8.9) | 82.0 (3.6) | 75.5 (8.7)
  Cohort 3, n=10, 3 | 76.5 (9.7) | 81.7 (11.0) | 77.7 (9.8)
  Cohort 4, n=10, 3 | 81.6 (6.1) | 76.7 (3.8) | 80.5 (5.9)
Sex/Gender, Customized [Number; unit: participants]
  Cohort 1, Female | 3 | 1 | 4
  Cohort 1, Male | 7 | 2 | 9
  Cohort 2, Female | 6 | 2 | 8
  Cohort 2, Male | 4 | 1 | 5
  Cohort 3, Female | 5 | 2 | 7
  Cohort 3, Male | 5 | 1 | 6
  Cohort 4, Female | 4 | 1 | 5
  Cohort 4, Male | 6 | 2 | 8
Best corrected visual acuity (BCVA) [Mean (Standard Deviation); unit: letters] — BCVA (with spectacles or other visual corrective devices) using Early Treatment Diabetic Retinopathy Study (ETDRS) testing was reported in letters read correctly out of 70 letters on the chart.
  letters
    Cohort 1, n=10, 3 | 63.4 (6.8) | 55.0 (8.7) | 61.5 (7.8)
    Cohort 2, n=10, 3 | 61.0 (11.8) | 64.3 (6.8) | 61.8 (10.7)
    Cohort 3, n=10, 3 | 60.2 (14.7) | 59.3 (5.1) | 60.0 (12.9)
    Cohort 4, n=10, 3 | 54.8 (14.2) | 48.7 (16.9) | 53.4 (14.4)
Central subfield thickness (CSFT) [Mean (Standard Deviation); unit: microns]
  Cohort 1, n=10, 3 | 535.1 (194.7) | 482.3 (104.3) | 522.9 (175.5)
  Cohort 2, n=10, 3 | 423.0 (95.5) | 405.7 (19.9) | 419.0 (83.5)
  Cohort 3, n=10, 3 | 479.1 (93.7) | 403.3 (67.7) | 461.6 (91.9)
  Cohort 4, n=10, 3 | 534.8 (123.4) | 573.3 (160.6) | 543.7 (126.5)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders Based on CSFT and BCVA Outcomes at Day 14 and Day 28
Description: A subject was considered a responder if at least 3 out of the following 4 criteria were fulfilled in comparison to baseline:
  * Greater than or equal to 4 letter gain in BCVA at Day 14
  * Greater than or equal to 4 letter gain in BCVA at Day 28
  * Greater than or equal to 80 micron decrease in CSFT at Day 14
  * Greater than or equal to 80 micron decrease in CSFT at Day 28. BCVA was measured by the number of letters read out of a possible 70 letters on the ETDRS chart. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 14, Day 28
Population: This analysis population includes all subjects who were randomized, received the initial injection or infusion, and had a baseline value and at least 1 postbaseline measurement for the period up to Day 28 for the primary efficacy variables (BCVA and/or CSFT). Here, "n" is the number of subjects in each arm group.
Measure: Number (90% Confidence Interval); unit: percentage of responders
Groups:
- Cohort 1: ESBA1008 solution Day 0 (1.2 mg) and Day 28 (6 mg), or Ranibizumab Day 0 and Day 28, based on randomization
- Cohort 2: ESBA1008 solution Day 0 (1 mg) and Day 28 (6 mg), or Ranibizumab Day 0 and Day 28, based on randomization
- Cohort 3: ESBA1008 solution Day 0 (0.6 mg) and Day 28 (6 mg), or Ranibizumab Day 0 and Day 28, based on randomization
- Cohort 4: ESBA1008 solution Day 0 (0.5 mg) and Day 28 (6 mg), or Ranibizumab Day 0 and Day 28, based on randomization
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 13 | 13 | 13 | 13
percentage of responders
  ESBA, n=10 | 70 [39.3 to 91.3] | 60 [30.4 to 85.0] | 80 [49.3 to 96.3] | 60 [30.4 to 85.0]
  LUCENTIS, n=3 | 100 [36.8 to 100.0] | 100 [36.8 to 100.0] | 33.3 [1.7 to 86.5] | 66.7 [13.5 to 98.3]

2. Secondary Outcome: Change From Baseline in BCVA, Cohort 1
Description: BCVA (with spectacles or other visual corrective devices) using ETDRS testing was reported in letters read correctly out of 70 letters on the chart. Improvement of BCVA was defined as an increase (gain) in letters read from the baseline assessment. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: This analysis population includes all subjects who were randomized, received the initial injection or infusion, and had a baseline value and at least 1 postbaseline measurement for the period up to Day 28 for the primary efficacy variables, with last observation carried forward (LOCF) imputation for missing values.
Measure: Mean (Standard Deviation); unit: letters
Groups:
- ESBA 1.2 mg INJ: All subjects treated with ESBA 1008 1.2 mg IVT injection
- LUCENTIS 0.5 mg INJ: All subjects treated with Ranibizumab 0.5 mg IVT injection
Arm/Group | ESBA 1.2 mg INJ | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
letters
  Day 7 | 4.5 (6.5) | 4.7 (7.4)
  Day 14 | 5.9 (6.1) | 6.3 (7.6)
  Day 28 | 7.7 (5.2) | 10.3 (6.1)
  Day 42 | 10.3 (4.9) | 8.3 (5.9)
  Day 56 | 11.1 (8.0) | 11.7 (5.5)

3. Secondary Outcome: Change From Baseline in BCVA, Cohort 2
Description: as for outcome 2
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: This analysis population includes all subjects who were randomized, received the initial injection or infusion, and had a baseline value and at least 1 postbaseline measurement for the period up to Day 28 for the primary efficacy variables, with LOCF imputation for missing values.
Measure: Mean (Standard Deviation); unit: letters
Groups:
- ESBA 1 mg INF: All subjects treated with ESBA 1008 1 mg IVT infusion
Arm/Group | ESBA 1 mg INF | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
letters
  Day 7 | 2.4 (6.2) | 7.0 (13.0)
  Day 14 | 4.8 (4.0) | 7.3 (10.4)
  Day 28 | 5.5 (6.0) | 10.3 (11.2)
  Day 42 | 8.1 (9.6) | 10.3 (11.0)
  Day 56 | 8.0 (7.3) | 10.7 (10.8)

4. Secondary Outcome: Change From Baseline in BCVA, Cohort 3
Description: as for outcome 2
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Groups:
- ESBA 0.6 mg INJ: All subjects treated with ESBA 1008 0.6 mg IVT injection
Arm/Group | ESBA 0.6 mg INJ | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
letters
  Day 7 | 10.3 (9.0) | 5.0 (4.6)
  Day 14 | 9.8 (12.0) | 7.3 (7.8)
  Day 28 | 13.5 (10.4) | 5.0 (6.9)
  Day 42 | 15.0 (10.1) | 6.0 (6.2)
  Day 56 | 13.7 (9.9) | 9.3 (1.5)

5. Secondary Outcome: Change From Baseline in BCVA, Cohort 4
Description: as for outcome 2
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: letters
Groups:
- ESBA 0.5 mg INF: All subjects treated with ESBA1008 0.5 mg IVT infusion
Arm/Group | ESBA 0.5 mg INF | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
letters
  Day 7 | 3.2 (6.0) | 9.3 (14.5)
  Day 14 | 7.1 (7.6) | 12.3 (11.8)
  Day 28 | 4.7 (3.8) | 11.7 (15.1)
  Day 42 | 6.6 (5.3) | 17.3 (17.9)
  Day 56 | 7.6 (7.1) | 18.7 (14.2)

6. Secondary Outcome: Change From Baseline in CSFT, Cohort 1
Description: CSFT was assessed by Spectral-Domain Optical Coherence Tomography (SD-OCT) and measured in microns. A decrease in CSFT indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Groups:
- ESBA 1.2 mg INJ: All subjects treated with ESBA1008 1.2 mg IVT injection
Arm/Group | ESBA 1.2 mg INJ | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
microns
  Day 7 | -114.0 (167.1) | -99.7 (16.3)
  Day 14 | -188.2 (122.0) | -130.3 (39.7)
  Day 28 | -182.0 (106.7) | -175.3 (71.8)
  Day 42 | -221.0 (156.3) | -183.7 (74.3)
  Day 56 | -226.3 (145.7) | -162.7 (68.6)

7. Secondary Outcome: Change From Baseline in CSFT, Cohort 2
Description: CSFT was assessed by SD-OCT and measured in microns. A decrease in CSFT indicates improvement. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Groups:
- ESBA 1 mg INF: All subjects treated with ESBA1008 1 mg IVT infusion
Arm/Group | ESBA 1 mg INF | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
microns
  Day 7 | -57.9 (38.1) | -87.7 (32.7)
  Day 14 | -96.5 (45.3) | -116.0 (19.7)
  Day 28 | -104.9 (44.2) | -142.3 (18.1)
  Day 42 | -133.1 (83.3) | -148.3 (26.0)
  Day 56 | -137.9 (73.9) | -155.0 (26.2)

8. Secondary Outcome: Change From Baseline in CSFT, Cohort 3
Description: as for outcome 7
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Groups:
- ESBA 0.6 mg INJ: All subjects treated with ESBA1008 0.6 mg IVT injection
Arm/Group | ESBA 0.6 mg INJ | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
microns
  Day 7 | -93.4 (50.1) | -54.0 (59.6)
  Day 14 | -126.8 (61.0) | -85.7 (87.4)
  Day 28 | -163.1 (74.4) | -104.0 (73.5)
  Day 42 | -194.4 (66.9) | -128.3 (73.8)
  Day 56 | -205.4 (78.6) | -108.7 (88.8)

9. Secondary Outcome: Change From Baseline in CSFT, Cohort 4
Description: as for outcome 7
Time Frame: Baseline, Day 7, Day 14, Day 28, Day 42, Day 56
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ESBA 0.5 mg INF | LUCENTIS 0.5 mg INJ
Number analyzed (Participants) | 10 | 3
microns
  Day 7 | -102.8 (111.1) | -105.3 (72.2)
  Day 14 | -119.9 (129.3) | -194.3 (148.9)
  Day 28 | -125.1 (143.6) | -187.3 (195.7)
  Day 42 | -184.2 (110.2) | -253.0 (181.2)
  Day 56 | -203.5 (105.8) | -213.7 (228.2)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of a subject's participation in the study (up to visit Day 56). Ocular adverse events are presented for both study eye and non-study eye. AEs were reported as pretreatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject administered study drug. AEs were obtained as solicited comments from subjects and as observations by the Investigator as outlined in the protocol.
Groups:
- Stage 1 ESBA 1.2 mg INJ: All subjects treated with ESBA1008 1.2 mg via injection
- Stage 1 ESBA 1 mg INF: All subjects treated with ESBA1008 1 mg via infusion
- Stage 1 LUCENTIS 0.5 mg INJ: All subjects treated with LUCENTIS via injection in Stage 1
- Stage 2 ESBA 0.6 mg INJ: All subjects treated with ESBA1008 0.6 mg via injection
- Stage 2 ESBA 0.5 mg INF: All subjects treated with ESBA1008 0.5 mg via infusion
- Stage 2 LUCENTIS 0.5 mg INJ: All subjects treated with LUCENTIS via injection in Stage 2
- Pretreatment: All subjects who consented to participate in the study prior to the initiation of study treatment
Arm/Group | Stage 1 ESBA 1.2 mg INJ | Stage 1 ESBA 1 mg INF | Stage 1 LUCENTIS 0.5 mg INJ | Stage 2 ESBA 0.6 mg INJ | Stage 2 ESBA 0.5 mg INF | Stage 2 LUCENTIS 0.5 mg INJ | Pretreatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/6 | 1/10 | 0/10 | 0/6 | 1/107
Other Adverse Events (participants affected / at risk) | 6/10 | 4/10 | 6/6 | 6/10 | 7/10 | 4/6 | 3/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 ESBA 1.2 mg INJ (N=10) | Stage 1 ESBA 1 mg INF (N=10) | Stage 1 LUCENTIS 0.5 mg INJ (N=6) | Stage 2 ESBA 0.6 mg INJ (N=10) | Stage 2 ESBA 0.5 mg INF (N=10) | Stage 2 LUCENTIS 0.5 mg INJ (N=6) | Pretreatment (N=107)
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 ESBA 1.2 mg INJ (N=10) | Stage 1 ESBA 1 mg INF (N=10) | Stage 1 LUCENTIS 0.5 mg INJ (N=6) | Stage 2 ESBA 0.6 mg INJ (N=10) | Stage 2 ESBA 0.5 mg INF (N=10) | Stage 2 LUCENTIS 0.5 mg INJ (N=6) | Pretreatment (N=107)
Androgen deficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Choroidal neovascularisation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Corneal epithelium defect (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eyelid pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retinal pigment epitheliopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Xanthopsia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Biopsy ear (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.